CLINICAL TRIAL: NCT00483444
Title: The Effect of Telephone Follow-Up on Outcome After Mild TBI
Brief Title: Telephone Follow-Up on Outcome After Mild Traumatic Brain Injury
Acronym: TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen Bell, Professor, Rehabilitative Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25091-G
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Brain Concussion
Keywords: Rehabilitation; Brain injuries; Directive counseling
MeSH Terms: conditions — Brain Concussion; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention): Control group were recruited in the emergency department after concussion and received standard care as directed by the ED physician and PCP.
- 1 (Experimental): Persons with concussion recruited in the emergency department received 5-6 scheduled telephone counseling calls focused on symptom management and self-management.
  Interventions: Behavioral: Scheduled telephone follow-up

INTERVENTIONS:
Behavioral: Scheduled telephone follow-up — Persons in the experimental group (group 1) received scheduled telephone counseling calls focused on symptom management and self-management skills.
  Arms: 1

SUMMARY:
The purpose of this study is to see whether providing education and counseling after a mild traumatic brain injury will help in preventing symptoms from becoming chronic over the first six months after injury.

DETAILED DESCRIPTION:
This study examines the effect of scheduled telephone calls on the outcome after mild traumatic brain injury (MTBI) or concussion. These calls offer subjects information, focused counseling, and referrals. MTBI is extremely common in the United States, numbering well over a million cases per year. Although recovery for most is quite good, 10-20% of persons have persisting symptoms that affect employment, quality of life, and health care expenses. We are examining one means to decrease persisting symptoms by offering early, consistent intervention before symptoms become persistent.

The subjects are enrolled in the emergency departments (ED) of the hospital and receive the baseline assessment while still in the ED. Subjects are randomly assigned to two groups: Group 1 standard care and Group 2 standard care, toll-free telephone number, and scheduled telephone calls for follow-up at 1-2 days, 2, 4, 8, and 12 weeks after injury. All subjects are contacted again at 6 months for an outcome assessment that is done over the telephone.

On the telephone, subjects are asked about current problems, and are given both information about recovery from MTBI and some counseling on dealing with symptoms or other complaints. They are also given community resources to obtain assistance if needed. Telephone call are reviewed by supervisors (physician and psychologist) for adherence to protocol and for training purposes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis consistent with mild traumatic brain injury
* Glasgow Coma Scale score 13-15
* Loss of consciousness less than or = to 30 minutes
* Any period of alteration of consciousness or post-traumatic amnesia
* age between 16 and 80
* permanent address
* ability to communicate in English

Exclusion Criteria:

* hospitalization within previous year for traumatic brain injury
* prior or current diagnosis of central nervous system or major psychiatric disorder
* Intoxication sufficient enough to cloud the diagnosis of mild TBI
* current alcohol dependence

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2003-10 (Actual); Primary Completion 2006-02 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Measure: two composite measures - post-traumatic symptoms that develop or worsen after the injury - general health status | Six months

SECONDARY OUTCOMES:
1. Improvement of functional level, emotional status, community activities, and perceived quality of life (SF-12 Health Survey, Patient Health Questionnaire - Depression and Anxiety Scales, Community Integration Scale, Perceived Quality of Life) | Six months
Assess the effectiveness of this intervention in subgroups defined by gender or race. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R Bell, M.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Bell KR, Hoffman JM, Temkin NR, Powell JM, Fraser RT, Esselman PC, Barber JK, Dikmen S. The effect of telephone counselling on reducing post-traumatic symptoms after mild traumatic brain injury: a randomised trial. J Neurol Neurosurg Psychiatry. 2008 Nov;79(11):1275-81. doi: 10.1136/jnnp.2007.141762. Epub 2008 May 9. PMID 18469027
- [Result] Hoffman JM, Dikmen S, Temkin N, Bell KR. Development of posttraumatic stress disorder after mild traumatic brain injury. Arch Phys Med Rehabil. 2012 Feb;93(2):287-92. doi: 10.1016/j.apmr.2011.08.041. PMID 22289239
- [Result] Powell JM, Ferraro JV, Dikmen SS, Temkin NR, Bell KR. Accuracy of mild traumatic brain injury diagnosis. Arch Phys Med Rehabil. 2008 Aug;89(8):1550-5. doi: 10.1016/j.apmr.2007.12.035. Epub 2008 Jul 2. PMID 18597735